CLINICAL TRIAL: NCT04787562
Title: A PHASE 1, OPEN-LABEL STUDY TO EVALUATE THE PHARMACOKINETICS AND SAFETY OF XNW4107, IMIPENEM AND CILASTATIN ADMINISTERED CONCURRENTLY AS INTRAVENOUS INFUSION TO SUBJECTS WITH VARIOUS DEGREES OF RENAL FUNCTION
Brief Title: Pharmacokinetics of XNW4107 in Subjects With Various Degrees of Renal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Evopoint Biosciences Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: XNW4107-003
Record Dates: First submitted 2021-03-01; First posted 2021-03-08 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Bacterial Infections
MeSH Terms: conditions — Bacterial Infections | interventions — Imipenem; Cilastatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort 1: normal renal function (Experimental): Participants with an eGFR ≥ 90 mL/min/1.73m2 receive a single dose of XNW4107 250mg IV co-administered with imipenem 500mg /cilastatin 500mg
  Interventions: Drug: XNW4107, Imipenem/Cilastatin
- Cohort 2: Mild renal insufficiency (Experimental): Participants with an eGFR 60 to <90 mL/min/1.73m2 receive a single dose of XNW4107 250mg IV co-administered with imipenem 500mg /cilastatin 500mg
  Interventions: Drug: XNW4107, Imipenem/Cilastatin
- Cohort 3: Moderate renal insufficiency (Experimental): Participants with an eGFR 30 to <60 mL/min/1.73m2 receive a single dose of XNW4107 250mg IV co-administered with imipenem 500mg /cilastatin 500mg
  Interventions: Drug: XNW4107, Imipenem/Cilastatin
- Cohort 4: Severe renal insufficiency (Experimental): Participants with an eGFR 15 to <30 mL/min/1.73m2 receive a single dose of XNW4107 100mg IV co-administered with imipenem 200mg /cilastatin 200mg
  Interventions: Drug: XNW4107, Imipenem/Cilastatin
- Cohort 5: End-stage renal disease (ESRD) receiving hemodialysis (HD) therapy (Experimental): Participants with ESRD receiving HD therapy at least 3 times a week for at least 3 months prior to Screening visit receive a single dose of XNW4107 100mg IV co-administered with imipenem 200mg /cilastatin 200mg
  Interventions: Drug: XNW4107, Imipenem/Cilastatin

INTERVENTIONS:
Drug: XNW4107, Imipenem/Cilastatin — Drug: XNW4107 250mg IV over 60 minutes as a single dose
  Drug: Imipenem/Cilastatin 500mg/500mg IV over 60 minutes as a single dose
  Arms: Cohort 1: normal renal function
Drug: XNW4107, Imipenem/Cilastatin — Drug: XNW4107 250mg IV over 60 minutes as a single dose
  Drug: Imipenem/Cilastatin 500mg/500mg IV over 60 minutes as a single dose
  Arms: Cohort 2: Mild renal insufficiency
Drug: XNW4107, Imipenem/Cilastatin — Drug: XNW4107 250mg IV over 60 minutes as a single dose
  Drug: Imipenem/Cilastatin 500mg/500mg IV over 60 minutes as a single dose
  Arms: Cohort 3: Moderate renal insufficiency
Drug: XNW4107, Imipenem/Cilastatin — Drug: XNW4107 100mg IV over 60 minutes as a single dose
  Drug: Imipenem/Cilastatin 200mg/200mg IV over 60 minutes as a single dose
  Arms: Cohort 4: Severe renal insufficiency
Drug: XNW4107, Imipenem/Cilastatin — Drug: XNW4107 100mg IV over 60 minutes as a single dose
  Drug: Imipenem/Cilastatin 200mg/200mg IV over 60 minutes as a single dose
  Arms: Cohort 5: End-stage renal disease (ESRD) receiving hemodialysis (HD) therapy

SUMMARY:
This is a Phase 1, open-label study to assess the PK, safety and tolerability of XNW4107, imipenem and cilastatin administered by 60-minute (60-min) IV infusion to adults with various degrees of renal insufficiency as compared to subjects with normal renal function.

ELIGIBILITY:
Inclusion Criteria:

* 1. Adult males or females, 18 years of age or older.

  2. BMI ≥ 18.5 and ≤ 39.9 (kg/m²) and weight between 50.0 and 130.0 kg (inclusive).

  3. Medically healthy (Cohort 1 only) or medically stable without clinically significant acute or chronic illness (Cohorts 2-5) that may impact the assessment of PK and safety.

  4. Normal renal function with eGFR ≥90 mL/min/1.73m² (Cohort 1), or renal insufficiency with eGFR 60 to <90 mL/min/1.73m² (Cohort 2), 30 to <60 mL/min/1.73m² (Cohort 3), or 15 to <30 mL/min/1.73m² (Cohort 4), ESRD receiving HDs at least 3 times per week for at least 3 months at Screening (Cohort 5)

  5. Participants of reproductive potential (male or female) must be willing to use contraception.

  6. Ability and willingness to abstain from alcohol, caffeine, xanthine-containing beverages or food or product containing any of these from 48 hours prior to study drug administration until discharge from the clinical unit.

Exclusion Criteria:

* 1. Any clinically significant medical history or abnormal findings upon physical examination, or clinical laboratory tests.

  2. Electrocardiogram (ECG) with QTcF interval duration equal or greater than 500 msec obtained at Screening or Check-In.

  3. Results for alanine aminotransferase (ALT), aspartate aminotransferase (AST) and bilirubin greater than 1.5 × the upper limit of normal (ULN) for the reference laboratory.

  4. History of chronic liver disease, cirrhosis, or biliary disease.

  5. History or presence of CNS disorders, seizures, or other CNS adverse reactions such as confusional states and myoclonic activity.

  6. Positive testing for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) at Screening.

  7. Close contact with anyone who tested positive for SARS-CoV-2 infection, or presence of symptoms associated with SARS-CoV-2 infection at Screening or Check-in, or within 14 days prior to Screening.

  8. Recent history (within 6 months) of known or suspected Clostridium difficile infection.

  9. Positive testing for HIV Ab, HBsAg or HCV Ab.

  10. Recent history of substance or alcohol abuse within the previous year, or habitual use of tobacco or nicotine products or smoking within 3 months prior to Screening.

  11. Positive drug screen and alcohol testing at Screening or Check-in.

  12. For subjects with normal renal function (Cohort 1), the use of any over-the-counter (OTC) medications within 7 days prior to study drug administration or use of prescription medications including nonsteroidal anti-inflammatory drugs, health supplements, and herbal remedies taken within 13 days prior to study drug administration.

  13. For subjects with renal impairment (Cohorts 2-5), the use of prohibited concomitant medication with the exception of those essential for the management of renal impairment and other concomitant stable medical conditions as per the discretion of the Investigator.

  14. Use of probenecid or valproic acid within 30 days prior to study drug administration.

  15. Receipt of an investigational drug within 30 days or 5 half-lives prior to the first administration of study drug, whichever is longer.

  16. Known history of clinically significant hypersensitivity reaction or anaphylaxis to any medication, or history of clinically significant hypersensitivity to the study drug or any related drugs or to any of the excipients, or history of food intolerance.

  17. Donation of blood or plasma within 30 days prior to dosing, or loss of whole blood of more than 500 mL within 30 days prior to dosing, or receipt of a blood transfusion within 1 year of study enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2021-02-25 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Total body clearance (CL) of XNW4107, imipenem and cilastatin in subjects with various of Renal function. | From baseline to 48 hours post-dose
Apparent steady-state volume of distribution (Vss) of XNW4107, imipenem and cilastatin in subjects with various of Renal function. | From baseline to 48 hours post-dose
Area under the curve from time zero to infinity (AUC0-∞)of XNW4107, imipenem and cilastatin in subjects with various of Renal function. | From baseline to 48 hours post-dose
Maximum plasma concentration (Cmax) of XNW4107, imipenem and cilastatin in subjects with various of Renal function. | From baseline to 48 hours post-dose
Time to the maximum plasma concentration (Tmax) of XNW4107, imipenem and cilastatin in subjects with various of Renal function. | From baseline to 48 hours post-dose
The terminal elimination half-life (t1/2) of XNW4107, imipenem and cilastatin in subjects with various of Renal function. | From baseline to 48 hours post-dose

SECONDARY OUTCOMES:
Adverse event (include SAEs) will be assessed and categorized. | From baseline up to 10 days post-dose
  Safety and tolerability up to the last study visit as assessed by the percentage of treatment-emergent AEs [including serious adverse events (SAEs)] categorized by severity, relationship to study drug, system organ class (SOC), AE preferred term (PT), along with percentage of clinically significant changes from baseline in clinical laboratory values, physical examination, vital signs, and ECG parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Le, Study Chair — Evopoint Biosciences Inc.
Locations (2):
- United States (2):
  - Division of Clinical Pharmacology (DCP), University of Miami, Miami, Florida
  - Orlando Clinical Research Center (OCRC), Orlando, Florida

IPD SHARING:
Plan to Share IPD: No